CLINICAL TRIAL: NCT03915743
Title: The AIR Project - Advance Care Planning Individualised Approach and Research Project. A Single Center Randomized Controlled Trial
Brief Title: Advance Care Planning Individualised Approach and Research Projec
Acronym: AIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristoffer Marsaa, Head of section, senior consultant MD, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIR
Record Dates: First submitted 2019-01-27; First posted 2019-04-16 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Severe COPD
Keywords: Palliative care; Out-patient clinic; COPD symptom burden
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative care (Experimental): Specialized palliative care arm in a newly formed COPD outpatient clinic
  Interventions: Other: palliative care
- Usual care (No Intervention): Usual care in a standard pulmonary out-patient clinic. Treatment as described in national standards.

INTERVENTIONS:
Other: palliative care — complex and multi-faceted individualized palliative care
  Arms: Palliative care

SUMMARY:
The study will investigate the effect of a palliative approach in the out-patient management of patients with COPD.

DETAILED DESCRIPTION:
Randomised control trial. A total of 90 patients will be randomise 1:1 to either palliative intervention or standard care.

The intervention group will receive follow up in a newly established outpatient clinic for COPD in the specialized palliative united and the control group will receive standard follow up in the respiratory out-patient clinic.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of COPD by spirometry

  * Patients followed in Herlev and Gentofte hospitals' respiratory out-patient-clinics or admitted to Herlev or Gentofte hospital for acute exacerbation
  * 2 or more admissions for acute exacerbation of COPD within the last 12 months
  * CAT > 20
  * Cognitive and linguistic able to understand and give informed consent

Exclusion Criteria:

* • Expected remaining life time less than 6 months due to other disease than COPD e.g. active cancer

  * Participating in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in total Hospital and Anxiety Depression scale (HADS) at 6 months | baseline, 3 and 6 months
  questionnaire measuring anxiety and Depression in 2 subscales in this study we use the total value of the 2 subscales combined. The higher the number the worse the psychological impact. HADS total was a range from 0 to 24 where 0 is no psychological distress

SECONDARY OUTCOMES:
Change from Baseline EORTC QLQ-C15-PAL at 6 months | baseline, 3 and 6 months
  questionnaire, consists of 14 questions and a license audit goal from 1 to 7 where 7 is the best possible quality of life.For the first 14 questions about symptoms, the scale goes from 1 to 4 where 4 is the worst
Change from Baseline Life-Space Assessment (LSA) at 6 months | baseline, 3 and 6 months
  questionnaire,5 questions about where the patient has been in the last 4 weeks. Question 1 is other than bedroom and question 5 is out of his home town. In addition, questions are asked about how frequently and on the use of aids.finally the scales are converted to numerical value between 0 and 120 where 0 is worst and expresses that the patient is constant in bed
Change from Baseline copd assessment test (CAT) at 6 months | baseline, 3 and 6 months
  questionnaire. 8 items questionnaire where there should be between 0 and 5 where 5 is the worst. Together, this gives a total scale between 0 and 40 where 40 is worst

OTHER OUTCOMES:
Adherence at 6months | 6 months
  measured by inhaled medicine bought at the pharmacy. Data is gather from a national database
Change from Baseline Use of out-patient clinic at 6 months | baseline to 6 months
  number of out-patient clinic visits
Change from Baseline in admission frequency at 6 months | baseline to 6 month
  numbers of admissions in the study periode

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Ulrik Jensen, Phd MD, Study Director — pulmonary department Herlev and Gentofte Hospital; Torgny Wilcke Wilcke, phd MD, Study Director — pulmonary department Herlev and Gentofte Hospital; Janni Mendahl, APN, Study Director — Palliative unite Herlev and Gentofte Hospital; Charlotte Ulrik, Prof. MD DMSc, Study Director — Pulmonary department Hvidovre Hospital; Nina Godtfredsen, phd MD, Study Chair — Pulmonary department Hvidovre Hospital; Kristoffer Marså, MD, Principal Investigator — Palliative Unite Herlev and Gentofte Hospital
Locations (1):
- Herlev & Gentofte hoospital, Copenhagen, Herlev/ Reghion H, Denmark

IPD SHARING:
Plan to Share IPD: No